CLINICAL TRIAL: NCT01068340
Title: Retrospective Review of the Incidence of Early Small Bowel Obstruction in Patients Undergoing an Exploratory Laparotomy Following Trauma
Brief Title: Early Small Bowel Obstruction Following Laparotomy For Trauma
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Demetrios Demetriades, Chief of Division of Acute Care Surgery and Surgical Critical Care, University of Southern California
Other Study IDs: EPSBO_TRAUMA_2010
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Small Bowel Obstruction
Keywords: Adhesions; Small Bowel Obstruction; Ileus
MeSH Terms: conditions — Tissue Adhesions; Ileus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SBO Patients: Patients who develop small bowel obstruction requiring or not surgical intervention
- No SBO Patients: Patients who do not develop small bowel obstruction

SUMMARY:
The formation of intraperitoneal adhesion following abdominal surgery is accepted by clinicians as an inevitable consequence. More than 90% of patients undergoing a surgical procedure in the abdomen will develop intraperitoneal adesions. The incidence however, of small bowel obstruction (SBO) resulting form these adhesions is far lower. To date, it is unknown which risk factors predispose these patients to develop SBO. Several have been proposed, such as age, peritonitis, or surgery for small bowel injury resulting from gunshots. None of them however, has been widely accepted.

During the last 20 years the significant lifetime risks associated with this phenomenon and its impact on the quality of life of patients has been well recognized. In addition, the burden on healthcare resources due to complications caused by adhesions is increasing and medicolegal consequences are rapidly evolving.

Early SBO following laparotomy for trauma is a poorly described entity. A few retrospective, single institution studies with a low number of patients have tried to address this issue. However, these studies either included a subset of trauma patients, i.e. patients sustaining penetrating trauma,[4] or patients undergoing a negative or non-therapeutic laparotomy, or examined only the incidence of SBO requiring surgical intervention. In addition, recent data regarding this issue is lacking, especially after the implementation of the damage control concept and the other advances in trauma surgery.

The aim of this study is to define the incidence of early SBO following laparotomy for trauma and to examine possible risk factors associated with its development.

DETAILED DESCRIPTION:
This is a retrospective review of all trauma patients admitted to the Los Angeles County - University of Southern California (LAC+USC) Medical Center from January 2006 to June 2009 (3.5 years). The trauma registry will be utilized to identify patients >= 15 years old who underwent a laparotomy during the study period and survived > 72 hours. For patients meeting inclusion criteria, all imaging studies obtained within the hospital course will be reviewed to identify patients who developed early SBO. The rationale for utilizing imaging studies is that obtaining these studies for patients with high suspicion of SBO is standard practice to establish the diagnosis. The charts of these patients will subsequently be reviewed and data will be collected using a predefined data collecting form.

ELIGIBILITY:
Inclusion Criteria:

* Exploratory laparotomy
* Survival > 72 hours

Exclusion Criteria:

* No exploratory laparotomy
* Survival <= 72 hours

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing an exploratory laparotomy for trauma
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Small Bowel Obstruction not requiring surgical intervention | 30 days

SECONDARY OUTCOMES:
Ileus | 30 days
Hospital length of stay | 30 days
Intensive Care Unit length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios Demetriades, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County + University of Southern California Medical Center, Los Angeles, California, United States